CLINICAL TRIAL: NCT00981539
Title: Do Preoperative Enemas Prevent Complications in Vaginal Pelvic Reconstructive Surgery?
Brief Title: Will Cleaning the Bowel With an Enema Before Vaginal Prolapse Surgery Prevent Complications?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illinois Urogynecology, Ltd. (Other)
Responsible Party: Denise M. Elser, MD, Illinois Urogynecology, LTD
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IULTD-4747
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Colon Cleansing
Keywords: The focus of this study is to determine whether it is beneficial to administer enemas before surgery
MeSH Terms: interventions — Enema

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment : receives pre operative enema (Active Comparator): one arm will receive pre operative enema
  Interventions: Procedure: enema
- no enema (No Intervention): this group will not receive pre operative enema

INTERVENTIONS:
Procedure: enema — pre operative rectal enema
  one adult bottle to be used rectally the night before surgery
  Other Names: adult over the counter enema
  Arms: treatment : receives pre operative enema

SUMMARY:
Traditionally, many gynecologic surgeons have asked patients to perform a cleansing enema the night before a vaginal surgery done to repair pelvic organ prolapse (dropped bladder, dropped uterus). The belief is that there is then less or no stool present at the vaginal incision and less chance of infection of the wound by bowel bacteria. However, not all surgeons follow this practice. There is no evidence in the medical literature if one way is better than the other. In this study, patients scheduled for vaginal surgery to correct prolapse will be randomly assigned to perform an enema or not to perform an enema.

DETAILED DESCRIPTION:
The factors to be measured will be wound infection rates, and need to cleanse an incision of escaped stool.

ELIGIBILITY:
Inclusion Criteria:

* female, AND
* undergoing vaginal surgery for prolapse.

Exclusion Criteria:

* pregnant women,
* age younger than eighteen,
* male sex, OR
* concurrent abdominal surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
wound infection rate | 6 weeks post op

SECONDARY OUTCOMES:
rate of contamination of surgical field by stool during surgery | day of surgery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Illinois Urogynecology, LTD., Oak Lawn, Illinois
  - Illinois Urogynecology, LTD., Park Ridge, Illinois

REFERENCES:
- See also: Practice site — http://www.iultd.org